CLINICAL TRIAL: NCT02154789
Title: An Assessment of Intra-lesional 3% Polidocanol Solution in the Treatment of Digital Myxoid Cysts
Brief Title: An Assessment of Intra-lesional 3% Polidocanol Solution in the Treatment of Digital Myxoid Cyst
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Foundation for Skin Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-005338-39
Record Dates: First submitted 2014-05-15; First posted 2014-06-03 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Ganglion Cysts
MeSH Terms: conditions — Ganglion Cysts | interventions — Polidocanol; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- polidocanol (Experimental)
  Interventions: Drug: polidocanol
- cryotherapy (Active Comparator)
  Interventions: Procedure: cryotherapy
- infra-red coagulation (Active Comparator)
  Interventions: Procedure: infra-red coagulation

INTERVENTIONS:
Drug: polidocanol
  Arms: polidocanol
Procedure: infra-red coagulation
  Arms: infra-red coagulation
Procedure: cryotherapy
  Arms: cryotherapy

SUMMARY:
Digital myxoid cysts arise from degeneration in the connective tissue of the digit joint, usually the last joint of the finger or toe, often due to underlying joint arthritis. They may connect with the joint. Pressure from the cyst can result in deformity of the digit's nail and trauma to the cyst results in leakage of the fluid, representing a potential source of entry for infection. Cysts can be tender and interfere with the digit's function. A variety of treatments are available, from simple extrusion which is rarely successful, to more destructive cryotherapy, infra-red coagulation and formal excision under local anaesthetic. These latter three approaches can result in considerable scarring. Sclerosant injection of polidocanol in one small non-randomised trial has been reported to be a well tolerated efficacious treatment with minimal scarring and long-term resolution. Following a pilot study, the investigators aim to trial this treatment to assess efficacy in a larger population.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to dermatology in NHS Lothian or NHS Fife who have a visible Digital Myxoid Cyst affective the dital phalynx of the toes or fingers.
* The patient must have the ability to give informed consent

Exclusion Criteria:

* History of sensitivity to polidocanol or other sclerosants
* Age less than 18
* Inability to give informed consent
* Inability to report side effects experienced
* Cyst not clearly visible
* Cyst not fluid-filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
cyst resolution at 6 weeks | 6 weeks
  Is there a difference in the percentage of participants with cyst resolution at 6 weeks post treatment in those treated with polidocanol compared to those treated with the current conventional treatments of cryotherapy and infra-red coagulation?

SECONDARY OUTCOMES:
cyst resolution at 12 and 52 weeks | 1 year
  In those participants treated with polidocanol compared to cryotherapy and also compared to infra-red coagulation is there a difference in the percentage of participants with cyst resolution at 12 and 52 weeks post initial treatment
difference in scarring | 1 year
  In those participants treated with polidocanol compared to cryotherapy and also compared to infra-red coagulation is there a difference in clinically apparent scarring
pain scores on a visual analogue scale | 1 year
  In those participants treated with polidocanol compared to cryotherapy and also compared to infra-red coagulation is there a difference in procedure pain/discomfort
procedure satisfaction on a visual analogue scale | 1 year
  In those participants treated with polidocanol compared to cryotherapy and also compared to infra-red coagulation is there a difference in procedure satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Holme, MBChB, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Queen Margaret Hospital, Whitefield Road, Dunfermline, Fife
  - Department of Dermatology, Royal Infirmary, Edinburgh, Midlothian